CLINICAL TRIAL: NCT00691327
Title: Adjunct Study of Natrelle(TM) Cohesive Round Silicone-Filled Breast Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan Medical (Industry)
Responsible Party: Sponsor
Organization: Allergan (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: 910044
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2013-12

CONDITIONS: Breast Reconstruction
Keywords: Revision of augmentation or reconstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Primary reconstruction
  Interventions: Device: Natrelle(TM) Silicone-Filled Breast Implants
- 2 (Experimental): Revision-reconstruction
  Interventions: Device: Natrelle(TM) Silicone-Filled Breast Implants
- 3 (Experimental): Revision-augmentation
  Interventions: Device: Natrelle(TM) Silicone-Filled Breast Implants

INTERVENTIONS:
Device: Natrelle(TM) Silicone-Filled Breast Implants — Breast implant surgery

SUMMARY:
Safety and effectiveness of Natrelle™ Cohesive Round Silicone-Filled Breast Implants in women undergoing primary reconstruction or revision of existing breast implants.

ELIGIBILITY:
Inclusion Criteria:

* Females of any age for which breast reconstruction is considered appropriate (Patients under 18 years old require parental/legal guardian consent to participate.
* Females seeking revision augmentation or revision reconstruction, where problems exist
* Have any of the following conditions or situations present:
* Post mastectomy surgical removal of the breast for cancer or other disease;
* Post trauma or post surgery where there was total or partial removal of the breast resulting in significant deformity;
* Severe ptosis requiring reconstruction;
* Any congenital or acquired discrepancy in breast size such as to represent a significant physical deformity.
* Adequate tissue available to cover implants.
* Saline-filled implants are not an appropriate choice.

Exclusion Criteria:

* Advanced fibrocystic disease considered to be premalignant without accompanying subcutaneous mastectomy.
* Existing carcinoma of the breast, without mastectomy.
* Abscess of infection in the body at the time of enrollment.
* Pregnant or nursing.
* Have any disease, including uncontrolled diabetes, which is clinically known to impact wound healing ability.
* Show tissue characteristics which are clinically incompatible with mammaplasty.
* Have, or under treatment for any condition which, in the opinion of the surgeon, may constitute an unwarranted surgical risk.
* Are not willing to undergo further surgery for revision, if medically required.
* Diagnosis of lupus or scleroderma.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84329 (Actual)
Dates: Start 1997-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Reconstruction: Women who have undergone Breast Reconstruction
- Revision: Women who have undergone Revision of a Breast Augmentation or Reconstruction
Period: Overall Study
Arm/Group | Reconstruction | Revision
Started | 45055 | 39274
Completed | 42214 | 36766
Not Completed | 2841 | 2508

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reconstruction | Revision | Total
Number analyzed (Participants) | 45055 | 39274 | 84329
Age, Customized [Number; unit: participants]
  <=17 years | 115 | 4 | 119
  Between 18 and 69 years | 43304 | 37612 | 80916
  >=70 years | 1065 | 1039 | 2104
  Not provided | 571 | 619 | 1190
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45055 | 39274 | 84329
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Local Complications
Description: By patient risk of complications occurring in at least 5% of patients in 1 or more cohorts
Time Frame: 5 years
Population: All enrolled patients
Measure: Number (95% Confidence Interval); unit: Percentage by Patient
Arm/Group | Reconstruction | Revision
Number analyzed (Participants) | 45055 | 39274
Percentage by Patient
  Capsular Contracture | 15.0 [14.4 to 15.6] | 21.6 [20.8 to 22.3]
  Asymmetry | 11.1 [10.6 to 11.7] | 10.7 [10.1 to 11.2]
  Implant Palpability/Visibility | 7.1 [6.7 to 7.6] | 11.4 [10.9 to 12.1]
  Implant Malposition | 6.5 [6.1 to 6.9] | 7.1 [6.7 to 7.6]
  Wrinkling | 5.6 [5.2 to 6.0] | 8.9 [8.4 to 9.4]
  Breast Pain | 5.2 [4.8 to 5.5] | 6.6 [6.1 to 7.0]

2. Secondary Outcome: Satisfaction With Breast Implants as Determined by Patients and Physicians on a 5-point Scale
Description: Satisfaction score on a 5-point scale, where 1 is definitely dissatisfied and 5 is definitely satisfied
Time Frame: 5 years
Population: All patients who had a breast implant satisfaction rating
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Reconstruction | Revision
Number analyzed (Participants) | 7426 | 5691
Units on a scale
  Physician Satisfaction | 4.4 (0.9) | 4.3 (1.0)
  Patient Satisfaction | 4.4 (0.9) | 4.3 (1.0)

ADVERSE EVENTS:
Arm/Group | Reconstruction | Revision
Serious Adverse Events (participants affected / at risk) | 0/45055 | 0/39274
Other Adverse Events (participants affected / at risk) | 0/45055 | 0/39274

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.